CLINICAL TRIAL: NCT05428878
Title: Prediction of Pregnancy Constitutions and Pregnancy Slippery Pulse Using ANSWatch
Brief Title: Pulse and Constitution of Pregnant Women
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH110-REC2-144
Record Dates: First submitted 2022-06-13; First posted 2022-06-23 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Pulse Wave; Pregnancy
Keywords: pregnant women; pulse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant: pregnant women
  Interventions: Diagnostic Test: ANS Watch
- Non-pregnant: non-pregnant women
  Interventions: Diagnostic Test: ANS Watch

INTERVENTIONS:
Diagnostic Test: ANS Watch — 1. ANS Watch will be used to record the pulse waves
  2. Constitution questionnaire will be used to measure the constitution type
  Other Names: Constitution questionnaire

SUMMARY:
The present project plans to detect pregnant pulses using this portable ANS (autonomic nervous system) Watch connected to a laptop. One hundred pregnant women and 100 non-pregnant women will be recruited.

DETAILED DESCRIPTION:
ANS(autonomic nervous system) Watch has been developed as to detect pulse waves using a pressure detector. It is used to measured cardiovascular indices, including cardiac output, and vessel stiffness. ANSWatch is developed to apply to the prediction of traditional Chinese medicine (TCM) pulses, such as the wiry pulse. There are 28 types of pulses in TCM. Among them, the slippery pulse is the most commonly seen pulse in pregnant women. The present project plans to detect pregnant pulses using this portable ANSWatch connected to a laptop. One hundred pregnant women and 100 non-pregnant women will be recruited. After taking the indices of the subjects, a neural network is designed to provide the prediction for pregnancy constitution, pregnancy pulse and slippery pulse in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* nonpregnant females and singleton pregnant females aged 20 - 45 years;
* no estrogen, progesterone, or ovulation inducing medications were in the past six months

Exclusion Criteria:

* active heart disease, liver disease, kidney disease, or thyroid disease;
* any chronic disease which needs medication
* smoking, drug abuse, or alcohol abuse;
* psychiatric disorders or impaired cognitive function;
* taking Chinese medicine or western medicine in three months;
* Acute conditions currently, such as gastroenteritis, upper airway infection, acute attach of asthma, etc.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females aged 20-45 years with a pregnant condition or a non-pregnant condition.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Pulse waves | Day 1
  The indices of pulse waves measured by ANSWatch , a pulse wave machine(https://www.taiwanscientific.com.tw/%E5%BF%83%E5%BE%8B%E5%A4%A7%E5%B8%ABanswatch).
  A neural network is designed to provide the prediction for pregnancy pulse.

SECONDARY OUTCOMES:
Constitution | Day 1
  Nine constitutions will be measured using the "Nine constitution Questionnaire" (in Chinese). This questionnaire defines whether subjects have Yin-deficiency, Yang-deficiency, Qi-deficiency, Phlegm-dampness, Dampness-heat, Special dialesis, Blood-stasis, Qi-depression, and Neuter constitutions.
  The questionnaire is divided into several sections, each addressing different aspects of the subject's constitution. Within each section, there are 6 to 8 sub-questions, and responses are rated on a scale from 1 to 5, reflecting the intensity or frequency of the subject's experiences.Sum the scores from all sub-questions within the section to obtain the raw score,which is then transformed to a 0-100 scale.
  If the transformed score falls below 30, it suggests that the subject does not exhibit characteristics of this constitution.Scores between 30 and 40 indicate a tendency towards this constitution.Scores exceeding 40 indicate that the subject belongs to this constitution.

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Yu Su, M.D., Principal Investigator — China Medical University, China
Locations (1):
- Shan-Yu Su, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plans to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Sanghavi M, Rutherford JD. Cardiovascular physiology of pregnancy. Circulation. 2014 Sep 16;130(12):1003-8. doi: 10.1161/CIRCULATIONAHA.114.009029. No abstract available. PMID 25223771
- [Background] Zhang YL, Zheng YY, Ma ZC, Sun YN. Radial pulse transit time is an index of arterial stiffness. Hypertens Res. 2011 Jul;34(7):884-7. doi: 10.1038/hr.2011.41. Epub 2011 May 19. PMID 21593741
- [Background] Pollonini L, Padhye NS, Re R, Torricelli A, Simpson RJ, Dacso CC. Pulse transit time measured by photoplethysmography improves the accuracy of heart rate as a surrogate measure of cardiac output, stroke volume and oxygen uptake in response to graded exercise. Physiol Meas. 2015 May;36(5):911-24. doi: 10.1088/0967-3334/36/5/911. Epub 2015 Apr 9. PMID 25856085
- [Background] Khalil SF, Mohktar MS, Ibrahim F. The theory and fundamentals of bioimpedance analysis in clinical status monitoring and diagnosis of diseases. Sensors (Basel). 2014 Jun 19;14(6):10895-928. doi: 10.3390/s140610895. PMID 24949644